CLINICAL TRIAL: NCT01890863
Title: An Open-Label, Randomised, Two Treatment, Four-Way Cross-Over (Replicate Design), Two Sequence, Repeat Dose, Single Centre Study in Healthy Volunteers to Compare the Pharmacokinetics of Fluticasone Propionate/Salmeterol (100/50 mcg) Delivered Via the Low Airflow Resistance ROTAHALER Inhaler Relative to Fluticasone Propionate/Salmeterol (100/50 mcg) Delivered Via the DISKUS Inhaler
Brief Title: ROTAHALER Device Optimization Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200260
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: asthma; fluticasone propionate/salmeterol; PK equivalence; COPD; pharmacokinetics; fluticasone propionate/salmeterol in a capsule-based inhaler; fluticasone propionate/salmeterol in a multi-dose dry powder inhaler; Respiratory
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Subjects will receive treatment A and B in following sequence in four treatment periods (one treatment per period): ABBA, where treatment A is 7 doses of FSC (100/50 mcg) delivered via the Ddpi and treatment B is 7 doses of FSC (100/50mcg) delivered via the Rdpi. Subjects will be dosed twice daily for 3 days and once on the fourth day in the morning (a single inhalation of 100/50mcg per dose).
  Interventions: Drug: Fluticasone Propionate / Salmeterol Xinafoate DISKUS; Drug: Fluticasone Propionate / Salmeterol Xinafoate ROTACAP
- Sequence 2 (Experimental): Subjects will receive treatment A and B in following sequence in four treatment periods (one treatment per period): BAAB, where treatment A is 7 doses of FSC (100/50 mcg) delivered via the Ddpi and treatment B is 7 doses of FSC (100/50mcg) delivered via the Rdpi. Subjects will be dosed twice daily for 3 days and once on the fourth day in the morning (a single inhalation of 100/50mcg per dose).
  Interventions: Drug: Fluticasone Propionate / Salmeterol Xinafoate DISKUS; Drug: Fluticasone Propionate / Salmeterol Xinafoate ROTACAP

INTERVENTIONS:
Drug: Fluticasone Propionate / Salmeterol Xinafoate DISKUS — Fluticasone propionate and salmeterol xinafoate combination as a dry powder inhaler for oral inhalation with unit dose strength of 100/50 mcg (available in blister pack) administered via DISKUS (Ddpi) device.
Drug: Fluticasone Propionate / Salmeterol Xinafoate ROTACAP — Fluticasone propionate and salmeterol xinafoate combination as a dry powder inhaler for oral inhalation with unit dose strength of 100/50 mcg (available in blister pack) administered via ROTAHALER (Rdpi) device.

SUMMARY:
This study will compare the pharmacokinetic (PK) of Fluticasone Propionate/Salmeterol combination (FSC) 100/50 micrograms (mcg) delivered via the capsule-based inhaler (Rdpi) relative to FSC 100/50 mcg delivered via the multi-dose dry powder inhaler (Ddpi) to establish whether the Rdpi inhaler has exposure (in terms of fluticasone propionate area under time concentration curve [AUC] and Salmeterol maximum concentration [Cmax]) no greater than 1.2500 compared to the Ddpi, sufficient to allow progression to Phase 3. This study will enroll 36 healthy adult male and female subjects and each subject will be allocated to one of two sequences and will participate in four treatment periods, receiving each of the treatments twice.

ELIGIBILITY:
Inclusion Criteria

* Males and females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator determines that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body mass index within the range 18 to 35 kilograms/meter squared (m^2) (inclusive).
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy (for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records); or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone > 40 milli international unit/mililiter [mL] and estradiol < 40 picogram/mL [<147 picomoles/liter] is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

Child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotropin (hCG) test at screening or prior to dosing.

Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 2 days post-last dose.

OR has only same-sex partners, when this is her preferred and usual lifestyle.

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Alanine aminotransferase, alkaline phosphatase and bilirubin <= 1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 %).
* Based on single or averaged QT interval corrected (QTc) values of triplicate electrocardiograms (ECGs) obtained over a brief recording period: QT duration corrected for heart rate by Fridericia's formula (QTcF)<450 millisecond (msec), and QT duration corrected for heart rate by Bazett's formula (QTcB)<480 msec in subjects with Bundle Branch Block.

Exclusion Criteria

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. In Australia one unit (= standard drink) is equivalent to 10 grams of alcohol: 270 mL of full strength beer (4.8%), 375mL of mid strength beer (3.5%), 470 mL of light beer (2.7%), 250 mL pre-mix full strength spirit (5%), 100 mL of wine (13.5%) and 30 mL of spirit (40%)
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immuno virus antibody.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Composite of PK parameters of FSC delivered via the Rdpi relative to FSC delivered via the Ddpi | PK samples will be collected at pre-dose, 5 minutes (mins), 10 mins, 30 mins, 1, 2, 4, 8, 10, and 12 hours post dose on Day 4 of each treatment period.
  PK Parameters include: area under the plasma fluticasone propionate concentration-time curve over dosing interval (AUCtau), salmeterol maximum plasma concentration-time curve on the last day of each study treatment period (Cmax).

SECONDARY OUTCOMES:
Composite of PK parameters of FSC delivered via the Rdpi relative to FSC delivered via the Ddpi | PK samples will be collected at pre-dose, 5 minutes (mins), 10 mins, 30 mins, 1, 2, 4, 8, 10, and 12 hours post dose on Day 4 of each treatment period.
  PK Parameters include: area under the plasma salmeterol concentration-time curve over dosing interval (AUCtau), fluticasone propionate maximum plasma concentration-time curve on the last day of each study treatment period (Cmax), and fluticasone propionate and salmeterol time of occurence of Cmax (Tmax) on the last day of each treatment period (Day 4).
Number of participants with adverse events (AEs) as measure of safety and tolerability. | 35 days.
  AEs will be collected from the start of study treatment and until the follow-up contact.
Laboratory parameters as a measure of safety and tolerability. | 35 days
  Laboratory parameters include: hematology, clinical chemistry, urinalysis and additional parameters.
Vital sign measurement as measure of safety and tolerability. | 35 days.
  Vital parameters include: systolic blood pressure, diastolic blood pressure, and pulse rate.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 200260 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200260?search=study&search_terms=200260#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 200260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200260 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register